CLINICAL TRIAL: NCT00181987
Title: Open-Label Study of Concerta in the Treatment of ADHD in Youth and Adults With Bipolar I, Bipolar II, and Bipolar Spectrum Disorder
Brief Title: Concerta in the Treatment of ADHD in Youth and Adults With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD; Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002-P-001148
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: ADHD; Bipolar Disorder
Keywords: ADHD; bipolar disorder; children; Concerta
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Bipolar Disorder | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate HCl (Concerta)

SUMMARY:
The objective of this study is to investigate the safety and effectiveness of Concerta in the treatment of children (ages 5 to 17 years old) and adults (ages 18 to 55 years old) with Bipolar I, Bipolar II and Bipolar Spectrum Disorder and comorbid ADHD over 8 weeks. This study seeks to study the short-term effectiveness of a long acting formulation of methylphenidate (Concerta) in the treatment of children and adults with bipolar disorder and comorbid ADHD adequately stabilized on an acceptable and stable regimen of anti-mania agents.

DETAILED DESCRIPTION:
A leading source of difficulty in treating youth with Bipolar Disorder is its comorbidity with attention deficit hyperactivity disorder (ADHD). Systematic studies of children and adolescents show that rates of ADHD range from 60% to 90% in pediatric study participants with mania. These findings could not be accounted for by the overlapping symptoms of distractibility, talkativeness, and physical hyperactivity, suggesting that affected children may suffer from both disorders, which was also consistent with findings of familial co-transmission of these two conditions. Considering the well-documented morbidity and dysfunction associated with ADHD, a comprehensive treatment approach to the management of the bipolar child with comorbid ADHD requires the development of appropriate therapeutic strategies for the treatment ADHD symptoms.

The objective of this study is to investigate the safety and effectiveness of Concerta in the treatment of children (ages 5 to 17 years old) and adults (ages 18 to 55 years old) with Bipolar I, Bipolar II and Bipolar Spectrum Disorder and comorbid ADHD over 8 weeks. This study seeks to study the short-term effectiveness of a long acting formulation of methylphenidate (Concerta) in the treatment of children and adults with bipolar disorder and comorbid ADHD adequately stabilized on an acceptable and stable regimen of anti-mania agents.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 5-55 years of age.
2. Each subject, as well as the legal representative for children under the age of 18, must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
3. Each subject (and his/her authorized legal representative, if applicable) must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the study participant must sign an informed assent document.
4. Subjects must have a diagnosis of Bipolar I, Bipolar II, Bipolar NOS or sub-threshold Bipolar Disorder with a stable Young Mania Scale rating of < 15 for at least one month, a Depression CGI-Severity score < 3 (mildly ill), a score on the Hamilton Depression Rating Scale below 15 (mild range), and a comorbid diagnosis of ADHD according to the DSM-IV based on clinical assessment and confirmed by structured diagnostic interview (Kiddie Schedule of Affective Disorders or Structured Clinical Interview DSM-IV), subjects may not have expressed symptoms for past 20 years.
5. Subject must be able to participate in mandatory blood draws.
6. Subject must be able to swallow pills.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Serious, unstable illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease
3. Uncorrected hypothyroidism or hyperthyroidism.
4. History of severe allergies or multiple adverse drug reactions.
5. Non-febrile seizures without a clear and resolved etiology.
6. Leukopenia or history of leukopenia without a clear and resolved etiology.
7. Judged clinically to be at serious suicidal risk.
8. Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol
9. History of intolerance or non-responder to Concerta as determined by the principal investigator.

Treatment with nonreversible monoamine oxidase inhibitor within 2 weeks prior to initiation of study.

Current diagnosis of schizophrenia. 12. Diagnosis of any chronic motor or vocal tic, or Tourette's Syndrome.

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2002-08; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Scores on the Young Mania Rating Scale
CGI-ADHD
ADHD-RS

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States